CLINICAL TRIAL: NCT06459349
Title: Effects of Exteroceptive and Proprioceptive Sensory Stimulation Versus Sensorimotor Therapy on Spasticity, Motor Function and Activities of Daily Living in Patients With Stroke
Brief Title: Effects of Sensory Stimulation Versus Sensorimotor Therapy on Spasticity, Motor Function and Daily Activities in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0282
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Stroke, Ischemic; Proprioceptive Disorders; Sensory Defect
Keywords: Stroke, Ischemic; Proprioceptive Disorders; Sensory Defect
MeSH Terms: conditions — Ischemic Stroke; Somatosensory Disorders

STUDY DESIGN:
Intervention Model Description: Patients will be divided to group A (n=21) which will receive intervention exteroceptive and proprioceptive sensory stimulation and to group B (n=21) which will receive sensorimotor therapy for 50 minutes per session, 03 times a week, for 06 weeks .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exteroceptive and proprioceptive sensory stimulation (Experimental): Patients in this group will receive exteroceptive and proprioceptive sensory stimulation
  Interventions: Other: exteroceptive and proprioceptive sensory stimulation training
- sensorimotor therapy group (Active Comparator): Patients in this group will receive sensorimotor therapy
  Interventions: Other: sensorimotor therapy group

INTERVENTIONS:
Other: exteroceptive and proprioceptive sensory stimulation training — Patients in this group will receive intervention exteroceptive and proprioceptive sensory stimulation for 50 minutes per session, 03 times a week, for 06 weeks
  Arms: exteroceptive and proprioceptive sensory stimulation
Other: sensorimotor therapy group — Patients will receive sensorimotor therapy for 50 minutes per session, 03 times a week, for 06 weeks
  Arms: sensorimotor therapy group

SUMMARY:
To compare effects of exteroceptive and proprioceptive sensory stimulation versus sensorimotor therapy on spasticity, motor function and activities of daily living in patients with stroke

DETAILED DESCRIPTION:
It will be a randomized clinical trial in which total 42 stroke patients will be recruited through non probability convenience sampling techniques. Data will be collected from Gujranwala Medical College Teaching Hospital and Riphah Rehabilitation Center Lahore. The patients who are fulfilling the inclusion criteria will be randomly assigned to either group A (n=21) which will receive intervention exteroceptive and proprioceptive sensory stimulation or to group B (n=21) which will receive sensorimotor therapy for 50 minutes per session, 03 times a week, for 06 weeks. Baseline treatment will be given to both groups. Conventional therapy will be given for 20 minutes per session, 03 times a week, for 06 weeks. Data collection tools will be Fugl-Meyer Assessment, Modified Barthel Index and Modified Ashworth Scale.

ELIGIBILITY:
Inclusion Criteria:

* The patients with chronic stroke (6 months to 2 years)
* Patient 's muscular activity on Stage 3 or higher according to the Brunnstrom's stages of stroke recovery.
* Patients having Mini Mental State Examination score > 24

Exclusion Criteria:

* Significant musculoskeletal impairments (e.g., arthritis, joint contractures).
* Any other neurological disorders like multiple sclerosis, Parkinson 's disease.
* History of orthopaedic surgery.
* Unstable medical conditions (e.g., uncontrolled hypertension, cardiovascular disease).
* Severe visual or vestibular impairments.
* Lower limb prosthesis.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | 6 months
  Fugl-Meyer Assessment:
  It is designed to evaluate functional recovery after stroke and is based on the poststroke recovery sequence. The test evaluates 5 domains of upper limb, lower limb, balance, sensation, and range of motion in 155 items. The overall reliability was high (overall intraclass correlation coefficient = .96), and the intraclass correlation coefficients for the subsections of the assessment varied from .61 for pain to .97 for the upper extremity. Greater scores refer to improvement in limb functions
Modified Barthel Index: | 6 months
  Modified Barthel Index:
  It assesses the level of ability to perform daily activities. This questionnaire measures one's ability to perform different aspects of daily performance on a 0 to 100 scale, with higher scores indicating better performance. 0 to 20 scores are considered as complete dependency, 20 to 60 grades as severe dependency, 61 to 90 as moderate dependency, 91 to 99 as partial dependency and 100 as complete independence.
The Modified Ashworth Scale | 6 months
  The Modified Ashworth Scale is used to assess muscle spasticity. Spasticity using this scale, is the amount of muscle tone that scores between 0 and 4. Score 0 means no increase in tone; score
  1 slight increase in muscle tone, with little resistance at the end of the flexion range or extension of involved limb; +1 score slight increase in muscle tone, characterized by slightly resistance at less than half the flexion or extension of involved limb; score 2 significant increase in muscle tone in most limb range;, score 3 significant increase in passive muscle tone, movement is difficult; and score 4 limb involved in flexion or extension rigidity.

CONTACTS AND LOCATIONS:
Overall Officials: Zeest hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zlokovic BV, Gottesman RF, Bernstein KE, Seshadri S, McKee A, Snyder H, Greenberg SM, Yaffe K, Schaffer CB, Yuan C, Hughes TM, Daemen MJ, Williamson JD, Gonzalez HM, Schneider J, Wellington CL, Katusic ZS, Stoeckel L, Koenig JI, Corriveau RA, Fine L, Galis ZS, Reis J, Wright JD, Chen J. Vascular contributions to cognitive impairment and dementia (VCID): A report from the 2018 National Heart, Lung, and Blood Institute and National Institute of Neurological Disorders and Stroke Workshop. Alzheimers Dement. 2020 Dec;16(12):1714-1733. doi: 10.1002/alz.12157. Epub 2020 Oct 8. PMID 33030307
- [Background] Serrada I, Hordacre B, Hillier SL. Does Sensory Retraining Improve Sensation and Sensorimotor Function Following Stroke: A Systematic Review and Meta-Analysis. Front Neurosci. 2019 Apr 30;13:402. doi: 10.3389/fnins.2019.00402. eCollection 2019. PMID 31114472
- [Background] Kim KH, Jang SH. Effects of Task-Specific Training after Cognitive Sensorimotor Exercise on Proprioception, Spasticity, and Gait Speed in Stroke Patients: A Randomized Controlled Study. Medicina (Kaunas). 2021 Oct 13;57(10):1098. doi: 10.3390/medicina57101098. PMID 34684135